CLINICAL TRIAL: NCT06117046
Title: The Cardio-protective Effect of Cardiomyopeptidin on Myocardial Injury in ICU Patients With Non-organic Heart Disease: a Prospective, Single-blind, Randomized Controlled Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-2023-060
Record Dates: First submitted 2023-09-14; First posted 2023-11-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Injury; ICU

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiopeptidin (Experimental): Cardiopeptidin was administered intravenously once a day with 60mg of cardiopeptide for 3 days
  Interventions: Drug: Cardiopeptidin
- 50 ml of normal saline intravenous infusion (Placebo Comparator): 50 ml of normal saline intravenous infusion.
  Interventions: Drug: 50 ml of normal saline intravenous infusion

INTERVENTIONS:
Drug: Cardiopeptidin — Cardiopeptidin was administered intravenously once a day with cardiopeptidin for 3 days.The dosing regimen follows the recommended dosage of 1 mg/kg/day as outlined in the product manual, with doses calculated based on the ideal body weight.
  Arms: Cardiopeptidin
Drug: 50 ml of normal saline intravenous infusion — 50 ml of normal saline intravenous infusion
  Arms: 50 ml of normal saline intravenous infusion

SUMMARY:
The study was a single-center, randomized controlled pilot study. To explore the cardioprotective effect of cardiopeptidin on non-heart disease patients with severe cardiac injury by comparing whether cardiopeptidin was used.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. The high-sensitive troponin T index was higher than the normal value during ICU hospitalization
3. Obtain the informed consent of the subject or legal agent

Exclusion Criteria:

1. Patients who are expected to die within 48 hours of ICU admission
2. previous diagnosis of acute coronary syndrome, chronic cardiomyopathy, pulmonary heart disease, acute myocarditis, pericardial tamponade and other diseases that have been confirmed to cause myocardial injury
3. cardiopulmonary resuscitation and/or electrical defibrillation before admission
4. patients with acute ischemic stroke
5. patients with stage 5 chronic kidney disease
6. during pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events | On the day of enrollment, until 28 days.
  major adverse cardiac events

SECONDARY OUTCOMES:
28-day all-cause mortality | 28-day
  28-day all-cause mortality
90-day all-cause mortality | 90-day
  90-day all-cause mortality
Cardiac adverse events | In hospital, until the patient is discharged.
  Cardiac adverse events
LVEF | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  LVEF
APACHE II | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  APACHE II
Hypersensitive troponin T | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
MB | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  MB
NT-Pro BNP | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  NT-Pro BNP
LDH | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  LDH
α-HBDH | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  α-HBDH
CK | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  CK
CKMB | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  CKMB
Lac | On the day of enrollment, 1/4/7/14 days after enrollment，up to two weeks
  Lac

CONTACTS AND LOCATIONS:
Overall Officials: zhenhua zeng, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university Nanfang hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR